CLINICAL TRIAL: NCT05423197
Title: Phase II Study Evaluating Zr-Panitumumab for Assessment of Suspected Metastatic Lesions on 18F-FDG-PET/CT in Head and Neck Squamous Cell Carcinoma
Brief Title: 89Zr-Panitumumab for Assessment of Suspected Metastatic Lesions on 18F-FDG-PET/CT in HNSCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-63234; ENT0095 (Other: Stanford OnCore)
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Head-and-neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- panitumumab 30 mg (Active Comparator): Subjects will be given a 30mg of panitumumab
  Interventions: Drug: Panitumumab
- 89Zr-panitumumab IV (Experimental): Subjects will be given 89Zr-panitumumab IV
  Interventions: Drug: 89Zr-panitumumab IV

INTERVENTIONS:
Drug: 89Zr-panitumumab IV — Subjects will be given a bolus of 1.0 mCi (range 0.8 - 1.2 mCi) of 89Zr-panitumumab before undergoing further standard of care diagnostic evaluation of the lesions
  Arms: 89Zr-panitumumab IV
Drug: Panitumumab — Panitumumab 30mg will be given orally
  Arms: panitumumab 30 mg

SUMMARY:
The purpose of this study is to determine the diagnostic utility of 89Zr-panitumumab to identify metastatic lesion(s) in subjects with head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE(S):

- Determine the sensitivity and specificity of 89Zr-panitumumab for the detection of suspected metastatic lesions

SECONDARY OBJECTIVE(S):

- Compare sensitivity and specificity of 18F-FDG-PET/CT and 89Zr-panitumumab-PET/CT for detection of suspected metastatic lesions

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years.
* Biopsy confirmed diagnosis of squamous cell carcinoma of the head and neck.
* Subjects diagnosed with any T stage, any subsite within the head and neck. Subjects with recurrent disease or a new primary will be allowed.
* Must have standard of care 18F-FDG-PET/CT scan ≤ 30 days of Day 0 with suspected metastatic lesions.
* Have acceptable hematological status, coagulation status, kidney function, and liver function including the following clinical results:

  * Hemoglobin ≥ 9gm/dL
  * White blood cell count > 3000/mm3
  * Platelet count ≥ 100,000/mm3
  * Serum creatinine ≤ 1.5 times upper reference range
  * PTT = 11.5 - 14.4 seconds
  * INR = 0.9 - 1.2

Exclusion Criteria:

* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment
* History of infusion reactions to other monoclonal antibody therapies
* Pregnant or breastfeeding
* Magnesium or potassium lower than the normal institutional values
* Subjects receiving Class IA (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents
* Subjects with a history or evidence of interstitial pneumonitis or pulmonary fibrosis
* Severe renal disease or anuria
* Known hypersensitivity to deferoxamine or any of its components

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of 89Zr-panitumumab | Up to 1 year
  The total number of head and neck squamous cell carcinoma-involved incidental lesions will be determined and correlated to the radiologically suspicious lesions identified by 89Zr-panitumumab using PET/CT imaging.

SECONDARY OUTCOMES:
Sensitivity and Specificity 89Zr-panitumumab compared to standard of care 18F-FDG PET/CT imaging | Up to 1 year
  The total number of head and neck squamous cell carcinoma-involved incidental lesions will be determined and correlated to the radiologically suspicious lesions identified by 18F-FDG using PET/CT imaging. The specificity and sensitivity of 89Zr-panitumumab will be compared to the specificity and sensitivity of 18F-FDG for identification of metastatic lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Baik, MD, Principal Investigator — Stanford Cancer Institute
Locations (1):
- Stanford Cancer Institute, San Francisco, California, United States